CLINICAL TRIAL: NCT04191616
Title: An Open-label, Phase 2 Study Treating Subjects With First or Second Relapse of Multiple Myeloma With Carfilzomib, Pomalidomide, and Dexamethasone (KPd)
Brief Title: Study of Early Relapsed, Lenalidomide-refractory Subjects Eligible for Carfilzomib Triplet
Acronym: SELECT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20180117; 2019-001169-34 (EudraCT Number)
Record Dates: First submitted 2019-11-22; First posted 2019-12-10 (Actual); Results first posted 2023-11-08 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: Multiple Myeloma; RRMM; Open-label; First Relapse Multiple Myeloma; Second Relapse Multiple Myeloma; Refractory to Lenalidomide; Triplicate Treatment Regimen; Dexamethasone; Carfilzomib; Pomalidomide
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — carfilzomib; Dexamethasone; Calcium Dobesilate; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Carfilzomib combined with pomalidomide and dexamethasone (Experimental): Carfilzomib, pomalidomide, and dexamethasone (KPd)
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone; Drug: Pomalidomide

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib will be administered intravenously over 30 ± 5 minutes, on days 1, 8, and 15 (± 2 days) of each 28-day cycle for up to 12 cycles or progression. A dose of 20 mg/m^2 will be administered on day 1 of cycle 1. All subsequent doses will be 56 mg/m^2. The frequency of carfilzomib administration will be reduced to day 1 and 15 per cycle starting with cycle 13 and continued until progression or end of study.
  Other Names: Kyprolis
Drug: Dexamethasone — Dexamethasone will be administered at least 30 minutes, but no more than 4 hours prior to carfilzomib on days of carfilzomib administration. Dexamethasone will be administered at a dose of 40 mg on days 1, 8, 15, and 22 of each 28-day cycle up to progression during cycles 1 to 12. Dexamethasone will be administered at a dose of 20 mg on days 1 and 15 of each 28-day cycle up to progression during cycles 13 onward. For subjects more than or equal to 75 years of age, the dose will be 20 mg during cycles 1 through 12 and 10 mg from cycles 13 onward.
  Other Names: Decadron, Ozurdex, DexPak 6, 10, 13 Day, ReadySHarp, LoCort, Maxidex
Drug: Pomalidomide — Pomalidomide dose will be 4 mg per day orally on days 1 to 21 of each cycle until progression.
  Other Names: Pomalyst

SUMMARY:
A Study Evaluating Treatment of Multiple Myeloma with Carfilzomib in Combination with Pomalidomide and Dexamethasone

DETAILED DESCRIPTION:
An Open-label, Phase 2 Study Treating Subjects with First or Second Relapse of Multiple Myeloma with Carfilzomib, Pomalidomide, and Dexamethasone (KPd)

This trial is designed to estimate the efficacy of a carfilzomib-based triplet in first or second relapse of multiple myeloma for subjects refractory to lenalidomide. The study is an open-label, phase 2 trial. Subjects may receive treatment until progression.

Myeloma disease status will be monitored locally for response and progression per International Myeloma Working Group (IMWG) criteria (Kumar et al, 2016) every 28 ± 7 days from cycle 1 day 1 until confirmed progressive disease (PD), death, lost to follow-up, or withdrawal of full consent (whichever occurs first), regardless of cycle duration, dose delays or treatment discontinuation. Subjects with a suspected complete response (CR) or better will have a bone marrow for minimal residual disease (MRD) assessment at 12 and 24 months (± 4 weeks) from start of treatment (unless a MRD assessment was performed within 4 months before planned assessment).

Subjects who end study drug(s) without confirmed PD are required to complete disease response assessments and report new anti-myeloma treatment every 28 ± 7 days until first subsequent anti-myeloma treatment, death, lost to follow-up, withdrawal of full consent, confirmed PD, or end of study, whichever occurs first. Subjects who discontinue treatment and either start new anti-myeloma treatment or have PD will enter long-term follow-up every 12 weeks until death or end of study.

Approximately one-third of subjects enrolled in the study will be in first relapse and two-thirds in second relapse.

This study will enroll adults ≥ 18 years of age with first or second relapse multiple myeloma.

Eligible subjects will have relapsed multiple myeloma after receiving 1 or 2 prior lines of therapy.

Subjects must be refractory to lenalidomide. Subjects may not have received prior pomalidomide. Prior exposure to a proteasome inhibitor is allowed. Subjects previously exposed to carfilzomib must have responded with at least a partial response to carfilzomib, must not have discontinued carfilzomib due to toxicity, may not have relapsed while receiving or within 60 days of the last dose of carfilzomib, and must have at least a 6 month carfilzomib treatment-free interval since their last dose of carfilzomib.

Subjects must have measurable disease per IMWG consensus criteria, Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 2, and at least partial response to 1 line of therapy.

ELIGIBILITY:
Inclusion Criteria

* Subject has provided informed consent prior to initiation of any study specific activities or procedures.
* Male or female subjects age ≥ 18 years
* First or second relapse of multiple myeloma by IMWG criteria (subjects refractory to the most recent line of therapy, excluding carfilzomib, are eligible)
* Refractory to lenalidamide
* Measurable disease with at least 1 of the following assessed within 28 days prior to enrollment:

  * IgG multiple myeloma: serum monoclonal protein (M-protein) level ≥ 1.0 g/dL
  * IgA, IgD, IgE multiple myeloma: serum M-protein level ≥ 0.5 g/dL
  * urine M-protein ≥ 200 mg per 24 hours
  * in subjects without measurable serum or urine M-protein, serum-free light chain (SFLC) ≥ 100 mg/L (involved light chain) and an abnormal serum kappa lambda ratio
* Must have at least a PR to at least 1 line of prior therapy
* Prior therapy with proteasome inhibitors is allowed. Subjects receiving prior carfilzomib therapy must have achieved at least a PR, was not removed due to toxicity, did not relapse within 60 days from discontinuation of carfilzomib, and must have at least a 6 month carfilzomib treatment-free interval from their last dose of carfilzomib
* ECOG PS of 0 to 2

Exclusion Criteria

* Primary refractory multiple myeloma
* Waldenström macroglobulinemia
* Multiple myeloma of IgM subtype
* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Plasma cell leukemia ( greater than 2.0 × 109/L circulating plasma cells by differential). If automated differential shows ≥ 20% of other cells, obtain manual differential to identify other cells.
* Primary amyloidosis (patients with multiple myeloma with asymptomatic deposition of amyloid plaques found on biopsy would be eligible if all other criteria are met)
* Previous diagnosis of amyloidosis associated with myeloma
* Myelodysplastic syndrome
* Toxicity requiring discontinuation of lenalidomide therapy
* Prior treatment with pomalidomide

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (46):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Rocky Mountain Cancer Centers Denver Midtown, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Affiliated Oncologists, LLC, Chicago Ridge, Illinois
  - Minnesota Oncology Hematology PA, Saint Paul, Minnesota
  - Oncology Hematology Care Incorporated, Cincinnati, Ohio
  - Texas Oncology - Austin Midtown, Austin, Texas
  - United States Oncology Regulatory Affairs Corporate Office, Austin, Texas
  - US Oncology Research Investigational Products Center, Austin, Texas
  - Baylor Charles A Sammons Cancer Center at Dallas, Dallas, Texas
  - Texas Oncology, Fort Worth, Fort Worth, Texas
  - Texas Oncology- Tyler, Tyler, Texas
  - Blue Ridge Cancer Care, Roanoke, Virginia
- Denmark (4):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus Universitetshospital, Aarhus N
  - Sjaellands Universitetshospital, Roskilde
  - Vejle Sygehus, Vejle
- North Estonia Medical Centre, Tallinn, Estonia
- France (7):
  - CHU Grenoble Alpes, Grenoble
  - Centre Hospitalier Régional Universitaire de Lille - Hôpital Claude Huriez, Lille
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Centre Hospitalier Universitaire de Bordeaux - Hôpital Haut Lévêque, Pessac
  - Centre Hospitalier de Saint Quentin, Saint-Quentin
  - Clinique Sainte Anne, Strasbourg
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
- Germany (4):
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Asklepios Klinik Altona, Hamburg
  - Universitätsklinikum Münster, Münster
  - Universitatsklinikum Tubingen, Tübingen
- Greece (7):
  - University General Hospital of Evros-Alexandroupolis District, Alexandroupoli
  - General Hospital Evangelismos, Athens
  - Alexandra Hospital, Athens
  - University Hospital of Ioannina, Ioannina
  - General University Hospital of Patras Panagia i Voithia, Pátrai
  - Theagenion Cancer Hospital of Thessaloniki, Thessaloniki
  - General Hospital of Thessaloniki Georgios Papanikolaou, Thessaloniki
- Italy (5):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona, Ancona
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia
  - Azienda Unita Sanitaria Locale LE Presidio Ospedaliero Vito Fazzi Polo Oncologico Giovanni Paolo II, Lecce
  - Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino Ospedale Molinette, Torino
- Spain (5):
  - Hospital Clinico Universitario de Salamanca, Salamanca, Castille and León
  - Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Perrot A, Delimpasi S, Spanoudakis E, Frolund U, Belotti A, Oriol A, Moreau P, McFadden I, Xia Q, Arora M, Dimopoulos MA. An open-label phase 2 study treating patients with first or second relapse of multiple myeloma with carfilzomib, pomalidomide, and dexamethasone (KPd): SELECT study. Leuk Lymphoma. 2024 Jun;65(6):833-842. doi: 10.1080/10428194.2024.2322030. Epub 2024 Mar 18. PMID 38497533
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 25 study centers in Denmark, France, Germany, Greece, Italy, Spain, and the United States from 06 August 2020 to 01 October 2024.
Pre-assignment Details: Participants with relapsed multiple myeloma whose disease was refractory to lenalidomide were enrolled.
Groups:
- Carfilzomib With Pomalidomide and Dexamethasone (KPd): Carfilzomib was administered intravenously on days 1, 8, and 15 (± 2 days) of each 28-day cycle for up to 12 cycles or progression or end of study. A dose of 20 mg/m^2 was administered on day 1 of cycle 1; all subsequent doses were 56 mg/m^2. From cycle 13, the frequency of carfilzomib administration was reduced to days 1 and 15 (± 2 days) per cycle until progression or end of study.
  Dexamethasone was administered orally or intravenously at a dose of 40 mg on days 1, 8, 15, and 22 of each cycle during cycles 1 to 12, and at a dose of 20 mg on days 1 and 15 from cycle 13 until progression or end of study.
  Pomalidomide 4 mg was administered orally on days 1 to 21 of each cycle until progression or end of study.
Period: Pre-assignment Period
Arm/Group | Carfilzomib With Pomalidomide and Dexamethasone (KPd)
Started | 54
Completed | 52
Not Completed | 2
Not completed — Did not receive study treatment | 2
Period: Treatment Period
Arm/Group | Carfilzomib With Pomalidomide and Dexamethasone (KPd)
Started | 52
Received Carfilzomib | 52
Received Pomalidomide | 52
Received Dexamethasone | 52
Completed | 0
Not Completed | 52
Not completed — Death | 37
Not completed — Sponsor decision | 11
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: Baseline measures are presented for the safety analysis set which included participants who received at least 1 dose of carfilzomib.
Arm/Group | Carfilzomib With Pomalidomide and Dexamethasone (KPd)
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black or African American | 1
  White | 47
  Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) As Assessed by the Independent Review Committee (IRC)
Description: Overall response was defined as the best overall confirmed response of: Complete response (CR): Negative immunofixation on serum and urine, soft tissue plasmacytomas disappearance, < 5% plasma cells in bone marrow (BM). Stringent CR (sCR): CR and normal serum free light chain ratio and no clonal cells in BM. Very Good Partial Response (VGPR): Serum and urine M-protein detectable by immunofixation or ≥ 90% reduction in serum M-protein (urine M-protein level < 100 mg/24-h). PR: ≥ 50% reduction of serum M-protein and 24-h urinary M-protein by ≥ 90% or to < 200 mg/24-h. Assessment was by IRC per International Myeloma Working Group Uniform Response Criteria (IMWG-URC). The 90% confidence intervals were estimated using the Clopper-Pearson method (1994).
Time Frame: From day 1 cycle 1 until the primary analysis (PA) data cutoff (DCO); the mean duration of KPd treatment as of the DCO was 42.0 weeks
Population: The safety analysis set included all participants who received at least 1 dose of carfilzomib.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib With Pomalidomide and Dexamethasone (KPd)
Number analyzed (Participants) | 52
percentage of participants | 57.7 [45.4 to 69.3]

2. Secondary Outcome: Percentage of Participants With a Minimal Residual Disease Negative Complete Response (MRD[-]CR) as Assessed by the IRC
Description: The MRD[-]CR rate was defined as the percentage of participants who reached MRD[-]CR at the 12 month landmark (8- to 13-month window). MRD[-]CR was defined as the achievement of CR (including sCR or better) per IMWG-URC by IRC assessment and MRD[-] status at a sensitivity of 10^-5 using next-generation sequencing based method in the bone marrow. The 90% CIs were estimated using the Clopper-Pearson method (1994).
Time Frame: Day 1 cycle 1 to month 12 (8 to 13 month window)
Population: The safety analysis set included all participants who received at least 1 dose of carfilzomib. The analysis was pre-specified until PA DCO only.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Carfilzomib With Pomalidomide and Dexamethasone (KPd)
Number analyzed (Participants) | 52
percentage of participants | 3.8 [0.7 to 11.6]

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as events with onset on or after the administration of the first dose of any study treatment and within the end of study, or 30 days after the last dose of any study treatment, whichever one was earlier, excluding events reported after end of study date.
Time Frame: From the first dose of any study treatment until the end of study or 30 days after the last dose of any study treatment, whichever occured earlier; Median (min, max) was 8.5 (1.0, 46.6) months
Population: The safety analysis set included all participants who received at least 1 dose of carfilzomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib With Pomalidomide and Dexamethasone (KPd)
Number analyzed (Participants) | 52
Participants | 50

4. Secondary Outcome: Number of Participants Achieving MRD[-] Response
Description: MRD[-] response was defined as achievement of MRD[-] status using next generation sequencing (NGS) based method in the bone marrow at any time.
Time Frame: From day 1 cycle 1 until the end of study (EOS); the mean duration of KPd treatment as of the EOS was 55.3 weeks
Population: The safety analysis set included all participants who received at least 1 dose of carfilzomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib With Pomalidomide and Dexamethasone (KPd)
Number analyzed (Participants) | 52
Participants | 5

5. Secondary Outcome: Number of Participants With Sustained MRD[-]CR for at Least 12 Months as Assessed by the IRC
Description: MRD[-]CR at the 12 months landmark was defined as achievement of CR (including sCR or better) per IMWG-URC by IRC and MRD[-] status at a sensitivity of 10^-5 using NGS based method in the bone marrow at the 12 months landmark (from 8 months to 13 months window). Maintaining MRD[-]CR for at least 12 months (- 4 weeks) was considered as sustained.
Time Frame: Day 1 cycle 1 to month 12 (8 to 13 month window)
Population: The safety analysis set included all participants who received at least 1 dose of carfilzomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib With Pomalidomide and Dexamethasone (KPd)
Number analyzed (Participants) | 52
Participants | 0

6. Secondary Outcome: Number of Participants With Sustained MRD[-]CR at Month 24 as Assessed by the IRC
Description: Sustained MRD[-]CR at 24 months included participants that maintained MRD[-]CR for 12 months or more after achieving MRD[-]CR status at 12 months.
Time Frame: Day 1 cycle 1 to month 26 (19 to 26 month window)
Population: The safety analysis set included all participants who received at least 1 dose of carfilzomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib With Pomalidomide and Dexamethasone (KPd)
Number analyzed (Participants) | 52
Participants | 0

7. Secondary Outcome: Kaplan-Meier Estimate of Duration of Response as Assessed by the IRC
Description: Disease response and progression were determined using IMWG-URC. Durations were calculated for responders. Medians and percentiles were estimated using the Kaplan-Meier method. 90% CIs for medians and percentiles were estimated using the method by Klein and Moeschberger (1997) with log-log transformation.
Time Frame: From day 1 cycle 1 until the PA DCO; the mean duration of KPd treatment as of the DCO was 42.0 weeks
Population: The safety analysis set included all participants who received at least 1 dose of carfilzomib. Only participants who achieved a partial response or better were included in the analysis.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Carfilzomib With Pomalidomide and Dexamethasone (KPd)
Number analyzed (Participants) | 30
months | 20.3 [9.2 to NA] — Upper confidence interval (CI) is N/A because it was not estimable due to data structure. Not enough events occurred at later times for reliable upper CI to be calculated.

8. Secondary Outcome: Time to Response as Assessed by the IRC
Description: Durations were calculated for responders. Time to response was defined as the time from start of any study treatment date to the earliest date when confirmed sCR, CR, very good partial response (VGPR), or partial response (PR) was first achieved.
Time Frame: From day 1 cycle 1 until the PA DCO; the mean duration of KPd treatment as of the DCO was 42.0 weeks
Population: as for outcome 7
Measure: Median (Full Range); unit: months
Arm/Group | Carfilzomib With Pomalidomide and Dexamethasone (KPd)
Number analyzed (Participants) | 30
months | 1.0 [1 to 2]

9. Secondary Outcome: Kaplan-Meier Estimate of Progression Free Survival (PFS) as Assessed by the IRC
Description: PFS was defined as time from start of treatment until progression or death from any cause. Medians and percentiles were estimated using the Kaplan-Meier method by Klein and Moeschberger (1997). 90% CIs for medians were estimated using the method by Klein and Moeschberger (1997) with log-log transformation.
Time Frame: From day 1 cycle 1 until the PA DCO; the mean duration of KPd treatment as of the DCO was 42.0 weeks
Population: The safety analysis set included all participants who received at least 1 dose of carfilzomib.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Carfilzomib With Pomalidomide and Dexamethasone (KPd)
Number analyzed (Participants) | 52
months | 11.1 [6.5 to NA] — Upper confidence interval (CI) is N/A because it was not estimable due to data structure. Not enough events occurred at later times for reliable upper CI to be calculated.

10. Secondary Outcome: Kaplan-Meier Estimate of Overall Survival (OS)
Description: OS was defined as the time from the start of treatment until death from any cause. Medians and percentiles were estimated using the Kaplan-Meier method. 90% CIs for medians were estimated using the method by Klein and Moeschberger (1997) with log-log transformation.
Time Frame: From day 1 cycle 1 until the EOS; the mean duration of KPd treatment was 55.3 weeks.
Population: The safety analysis set included all participants who received at least 1 dose of carfilzomib.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Carfilzomib With Pomalidomide and Dexamethasone (KPd)
Number analyzed (Participants) | 52
months | 17.6 [11.2 to 23.5]

11. Secondary Outcome: Number of Participants With Best Overall Confirmed Response of CR or Better as Assessed by the IRC
Description: The number of safety analysis set participants whose best overall response was sCR or CR per IMWG-URC over the duration of the study.
Time Frame: From day 1 cycle 1 until the PA DCO; the mean duration of KPd treatment as of the DCO was 42.0 weeks
Population: The safety analysis set included all participants who received at least 1 dose of carfilzomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib With Pomalidomide and Dexamethasone (KPd)
Number analyzed (Participants) | 52
Participants | 3

ADVERSE EVENTS:
Time Frame: All-cause mortality: from enrollment until the end of study or death date, whichever occurs later; Median (min, max) time on study was 15.2 (0.0, 47.0) months. Adverse events: from the first dose of any study treatment until the end of study or 30 days after the last dose of any study treatment, whichever occurs earlier; Median (min, max) was 8.5 (1.0, 46.6) months
Description: All-cause mortality is reported for all participants enrolled in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Carfilzomib With Pomalidomide and Dexamethasone (KPd)
All-Cause Mortality (participants affected / at risk) | 37/54
Serious Adverse Events (participants affected / at risk) | 22/52
Other Adverse Events (participants affected / at risk) | 48/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib With Pomalidomide and Dexamethasone (KPd) (N=52)
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Left ventricular failure (Cardiac disorders) | 1
Pyrexia (General disorders) | 1
COVID-19 (Infections and infestations) | 2
COVID-19 pneumonia (Infections and infestations) | 2
Clostridium difficile infection (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Infection (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Confusional state (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Renal disorder (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Bronchitis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib With Pomalidomide and Dexamethasone (KPd) (N=52)
Anaemia (Blood and lymphatic system disorders) | 16
Leukopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 9
Fatigue (General disorders) | 12
Oedema peripheral (General disorders) | 11
Pyrexia (General disorders) | 8
COVID-19 (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 6
Platelet count decreased (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6
Paraesthesia (Nervous system disorders) | 5
Syncope (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 8
Hypertension (Vascular disorders) | 8
Lower respiratory tract infection (Infections and infestations) | 3
Respiratory tract infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT04191616/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/16/NCT04191616/SAP_001.pdf